CLINICAL TRIAL: NCT00902668
Title: A Phase II Study Using Lovastatin to Improve Cosmetic Outcome After Radiation Therapy for Breast Cancer
Brief Title: Lovastatin in Reducing Side Effects After Radiation Therapy in Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-12044; HM12044 (Other: VCU IRB); CDR0000642246 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-01188 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Radiation Toxicity
Keywords: radiation toxicity; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries; Breast Carcinoma In Situ | interventions — Lovastatin; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (lovastatin) (Experimental): Patients undergo 25-28 fractions of standard whole-breast irradiation followed by a boost to the tumor bed or 10 fractions of accelerated partial-breast irradiation with balloon brachytherapy BID over 5-10 days. Patients also receive lovastatin PO QD for 12 months beginning on day 1 of radiation therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lovastatin; Other: questionnaire administration; Procedure: adjuvant therapy; Radiation: accelerated partial breast irradiation; Radiation: external beam radiation therapy

INTERVENTIONS:
Drug: lovastatin
Other: questionnaire administration
Procedure: adjuvant therapy
Radiation: accelerated partial breast irradiation
Radiation: external beam radiation therapy

SUMMARY:
RATIONALE: Drugs, such as lovastatin, may protect normal cells from the side effects of radiation therapy.

PURPOSE: This phase II trial is studying how well lovastatin works in reducing side effects after radiation therapy in women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the incidence of good/excellent cosmetic outcome, as defined by the Harvard Scale, after radiotherapy in women treated with lovastatin, as compared to historical controls.

OUTLINE: Patients undergo standard external beam whole-breast irradiation and/or accelerated partial breast irradiation. Patients receive oral lovastatin once daily beginning on the first day of radiotherapy and continuing for 12 months in the absence of disease progression or unacceptable toxicity.

Patients complete a questionnaire, the Breast Cancer Treatment Outcome Scale, at baseline and then at 6 months, 12 months, and 3 years after completion of radiotherapy to assess cosmetic and functional outcomes.

After completion of radiotherapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of invasive or in situ epithelial cancer of the breast

  * Stage 0, I, or II (Tis, T1, or T2) disease
  * Unifocal disease (single focus that can be encompassed by breast-conserving surgery)
* Has undergone prior surgical resection of the primary lesion (lumpectomy) and axillary nodal evaluation (if invasive disease is present)

  * Negative surgical margins (≥ 1 mm)
* Planning to undergo radiotherapy with either standard external beam radiotherapy or accelerated partial breast irradiation (interstitial or balloon brachytherapy)
* No Paget disease of the nipple
* No evidence of distant metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Karnofsky performance status 70-100%
* Transaminases < 3 times upper limit of normal (ULN)
* Creatine kinase < 5 times ULN
* Creatinine clearance ≥ 30 mL/min
* Negative pregnancy test
* No active liver or muscle disease
* No history of collagen vascular disease (e.g., systemic lupus erythematosus, scleroderma, or dermatomyositis)
* History of prior malignancy allowed provided life expectancy is ≥ 4 years
* No major medical or psychiatric illness that, in the investigator's opinion, would prevent completion of study treatment or interfere with follow-up
* No contraindication to an HMG-coA-reductase inhibitor

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the breast, lung, or mediastinum

  * Prior radiotherapy to the contralateral breast allowed
* No chemotherapy for ≥ 2 weeks prior to, during, and for ≥ 2 weeks after completion of radiotherapy
* No concurrent cytochrome P450 3A4 inhibitors
* Concurrent HMG-coA-reductase inhibitor allowed provided patient is able to switch to 20 mg of lovastatin per day
* Concurrent tamoxifen or an aromatase inhibitor allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie W. Cuttino, MD, Principal Investigator — Massey Cancer Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open to accrual from 4/21/09 to 3/2/10. Patients were recruited from radiation oncology clinics.
Pre-assignment Details: Patients can be registered only after pretreatment evaluation is completed and eligibility criteria are met. Protocol treatment begins on the first day of external beam radiation therapy or on the first day of brachytherapy and continues for 12 months.
Period: Overall Study
Arm/Group | Supportive Care (Lovastatin)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Protocol stopped due to slow accrual. | 3

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Lovastatin)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Good/Excellent Cosmetic Outcome During the First 5 Years After Radiotherapy
Description: Proportion of good or excellent cosmetic outcomes, assessed using the Harvard Cosmesis Scale
Time Frame: during the first 5 years after treatment
Population: Due to slow accrual the study was closed to accrual and all 3 participants were terminated. No data was analyzed.
Arm/Group | Supportive Care (Lovastatin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline to Off Study. 7 months or less
Arm/Group | Supportive Care (Lovastatin)
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Lovastatin) (N=3)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Infection with unknown ANC - Vagina (Infections and infestations) | 1 (2)
Fibrosis-cosmesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Breast (General disorders) | 1 (2)
Pain - Extremity-limb (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to no subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No